CLINICAL TRIAL: NCT06493279
Title: A Single-arm, Open-label, Phase I Clinical Study to Evaluate the Safety and Efficacy of a Single Intrathecal Injection of RJK002 in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Evaluate the Safety and Efficacy of Intrathecal Injection of RJK002 in Patients With Amyotrophic Lateral Sclerosis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RJK Biopharma Ltd (Industry)
Collaborators: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJK002-0001-R
Record Dates: First submitted 2024-07-02; First posted 2024-07-09 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Amyotrophic Lateral Sclerosis Als
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RJK002 Intrathecal injection (Experimental): Eligible subjects will receive a single intrathecal administration of investigational product. 9 subjects will be involved in 3 doses cohort from low to high: 6E13 vg/person, 1.2E14 vg/person, and 2.4E14 vg/person, 3 subjects for each cohort.
  Interventions: Drug: RJK002 Intrathecal injection

INTERVENTIONS:
Drug: RJK002 Intrathecal injection — Eligible subjects will receive a single intrathecal administration of investigational product with dose 3E13vg (3ml), 6E13vg(6ml), and 1.2E14 vg(12ml) per person sequentially.

SUMMARY:
The goal of the study aims to evaluate the safety and tolerability of a single intrathecal injection of RJK002 in subjects with amyotrophic lateral sclerosis (ALS), and to determine the recommended Phase II dose (RP2D).

ELIGIBILITY:
Main Inclusion Criteria:

1. Female or male subjects who are ≥ 18 years of age at screening;
2. Patients with a diagnosis consistent with clinically or laboratory-supported possible, probable, or definite sporadic or familial ALSALS in accordance with Revised EI Escorial diagnostic criteria published by the World Federation of Neurology (WFN);
3. The duration of the disease from the first symptom (any ALS symptom) prior to the screening visit must be less than 2 years (inclusive);
4. The Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) score ≥30 during the screening period, and the three respiratory scores (dyspnea, upright respiration, and respiratory insufficiency) must be ≥3;
5. The forced vital capacity (FVC) of predicted during the screening period is ≥70% at screening;
6. Body mass index (BMI) greater than 18 kg/m2 at screening;

Main Exclusion Criteria:

1. Subjects with other neurological diseases similar to ALS that affect the evaluation of drug efficacy, such as cervical spondylotic myelopathy, syringomyelia, spinal cord and brain stem tumors, hirayama disease, multifocal motor neuropathy, multiple sclerosis, Guillain-Barre syndrome, Parkinson's disease and dementia;
2. Patients with a diagnosis consistent with clinically or laboratory-supported possible, probable, or definite sporadic or familial ALSALS in accordance with Revised EI Escorial diagnostic criteria published by the World Federation of Neurology (WFN);
3. Subjects who refuse to take food and medication by nasal feeding tube during the study period due to swallowing dysfunction;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
incidence of adverse events (AEs)/serious adverse events (SAEs) | Each visit within 5 years after administration
Dose limiting toxicities (DLT) | 28 days after administration
  Measured as any drug-related serious adverse event that meet DLT standard. If a dose has less than 33% DLTs it will be considered tolerable.

SECONDARY OUTCOMES:
Change in the ALS Functional Rating Scale-revised (ALSFRSr) Score | 28 days, 56 days, 84 days, 6 months, 12months, 18 months after administration
  The ALSFRSr, a questionnaire-based scale assessing daily living function ranging from 48 (best score) to 0 (worst), was administered to the patient, or to a proxy if the patient could not communicate effectively. Decline was defined as ALSFRSr at baseline minus ALSFRSr at month 9. A positive value indicates worsening.

OTHER OUTCOMES:
change of concentration of neurofilament light chain (NFL) in blood and CSF | 84 days, 6 months, 12months, 18 months after administration

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Part of the data are planed to share on Oct 2025, Oct 2026, and Sep 2032.
Supporting Information: CSR